CLINICAL TRIAL: NCT06864351
Title: Prospective Evaluation of OptiThyDose, a Mathematical Model for Calculating Appropriate Dose Ranges in Children With Thyroid Diseases
Brief Title: Prospective Evaluation of OptiThyDose
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital Basel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-00046; ks21Szinnai
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Thyroid Diseases; Congenital Hypothyroidism; Graves Disease
MeSH Terms: conditions — Thyroid Diseases; Congenital Hypothyroidism; Graves Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group w/ Congenital Hypothyroidism (No Intervention): Patients with Congenital Hypothyroidism receiving routine levothyroxine (LT4) treatment
- OptiThyDose w/ Congenital Hypothyroidism (Experimental): Patients with Congenital Hypothyroidism receiving routine levothyroxine (LT4) treatment
  Interventions: Other: OptiThyDose
- Control group w/ Graves' Disease (No Intervention): Patients with Graves' Disease receiving routine carbimazole (CMZ) or methimazole (MMZ) treatment
- OptiThyDose w/ Graves' Disease (Experimental): Patients with Graves' Disease receiving routine carbimazole (CMZ) or methimazole (MMZ) treatment
  Interventions: Other: OptiThyDose

INTERVENTIONS:
Other: OptiThyDose — OptiThyDose is an iterative mathematical model applied at each patient visit, consisting of three components: (i) a disease-specific pharmacometrics (PMX) model, (ii) an empirical Bayesian estimation (EBE) component, and (iii) an optimal control theory (OCT) component. It calculates the optimal LT4 or CMZ/MMZ dose to maintain Free Thyroxine (FT4) levels within the upper half of the age-specific reference range, integrating past clinical and lab data.
  Dosing follows international guidelines, with physicians able to consult OptiThyDose for individualized dosing within recommended ranges. At each outpatient visit, the physician can either (A) prescribe a dose within OptiThyDose's suggested range or (B) choose a dose based on personal experience.
  Arms: OptiThyDose w/ Congenital Hypothyroidism; OptiThyDose w/ Graves' Disease

SUMMARY:
The aim of this multicentric, randomised, two-arms and single-blinded clinical trial is to prospectively evaluate OptiThyDose for Congenital hypothyroidism (CH) and Graves' disease (GD).

DETAILED DESCRIPTION:
Thyroid diseases can affect people from birth to adulthood, ith some being present at birth (congenital) and others developing later in life (acquired). These diseases need to be treated quickly and properly because if left untreated, they can impact brain development, thinking abilities, growth, puberty, and other important body functions. However, treating thyroid diseases in children can be challenging, as it's important to avoid both under- and overdosing.

Algorithms that help determine the best individual dose for children with thyroid diseases could reduce the risk of long-term problems, like impaired thinking and growth. This is especially important because cases of thyroid diseases in children are increasing worldwide.

OptiThyDose is a new mathematical model developed to help doctors find the right dose for children with thyroid diseases.

The primary goal of this multicentric, randomised, two-arms and single-blinded study is to test how well OptiThyDose works for children with two types of thyroid diseases: Congenital Hypothyroidism (CH) and Graves' Disease (GD).

If proven effective, OptiThyDose could help ensure more accurate dosing of thyroid medications, leading to better hormone control, fewer side effects, and improved health outcomes in children with Congenital Hypothyroidism (CH) and Graves' Disease (GD).

ELIGIBILITY:
Inclusion Criteria:

Congenital hypothyroidism (CH)

* Newborns with pathological neonatal screening and confirmation of an increased Thyrotropin (TSH) level in an independent venous blood sample

Graves' disease (GD)

* Children until 18 years with new diagnosis of GD, recurrence of GD, or insufficiently controlled GD under CMZ/MMZ during follow-up according to:

  * Pathological lab values (suppressed TSH, increased thyroid hormone levels, positive Anti-TSH-receptor antibodies)
  * Typical clinical picture, if present (goitre, tachycardia, palpitations, weight loss, hyperphagia, altered mood)

CH and GD

* The study participant must be accessible for scheduled visits, treatment and follow-up.
* Signed Informed Consent form (ICF) obtained prior to any study related procedure. Written IC for study participation must be signed and dated by the patient and/or his/her legal representative(s) in accordance with national legal requirements

Exclusion Criteria:

CH and GD

* Exclusion of newborns from mothers with GD
* Exclusion of patients in case of a life-threatening event

GD

* Exclusion of children with known other aetiologies of hyperthyroidism than GD without elevated Anti-TSH-receptor antibodies e.g.:

  * known toxic thyroid nodules proven by ultrasound/scintigraphy
  * known amiodarone induced hyperthyroidism
  * known McCune Albright syndrome (based on clinical, laboratory, and genetic diagnosis) associated hyperthyroidism
  * known genetically proven hyperthyroidism caused by activating mutations of the TSH receptor gene

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Serum Free Thyroxine (FT4) value | 90 days post treatment start
  The serum Free Thyroxine (FT4) values is evaluated. FT4, interpreted according to the age of patients, is used in clinical routine as marker of the adequacy of:
  * Thyroid hormone substitution with LT4 of insufficient thyroid function in patients with CH (low FT4 levels in case of under-dosing of LT4, high FT4 levels in case of over-dosing of LT4)
  * Suppression of overactive thyroid function with CMZ/MMZ in patients with GD (low FT4 levels in case of over-dosing of CMZ/MMZ, high FT4 levels in case of under-dosing of CMZ/MMZ)

SECONDARY OUTCOMES:
Proportion of Thyroid Hormone Levels Within Target Range | 90 days post treatment start and up to 1 year post treatment start
  The proportion of serum Thyroid Hormone Levels (FT4, TSH, FT3, T3, and T4) that fall within the upper half of the local laboratory reference range at the time point closest to 90 days after treatment initiation.
Deviations from Local Laboratory Reference Ranges for Thyroid Hormones | Up to 1 year post treatment start
  Assessment of deviations in serum thyroid hormone levels (time point, magnitude of elevation, area under the curve (AUC), and fold change) when exceeding the upper or falling below the lower limit of the respective local laboratory reference range.
Number of clinical visits | Up to 1 year post treatment start
  The number of routine clinical visits as required.
Disease-related adverse events | Up to 1 year post treatment start
  Assessment of Disease-related adverse events (number and type) occurring during the study period.
Average daily dose of administered drugs per kg | Up to 1 year post treatment start
  Assessment of the average daily dose per kilogram of administered drugs (LT4 or CMZ/MMZ) throughout the study period.

OTHER OUTCOMES:
Heart Rate | Up to 1 year post treatment start
  Assessment of heart rate measured both on-site and with a wearable device, at or between clinical visits, during the study period
Overall Treatment Costs | Up to 1 year post treatment start
  Evaluation of overall treatment costs (e.g. expenses based on the number of consultations and costs for laboratory measurements) from a health economic perspective during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Gabor Szinnai, Prof. MD, PhD, Principal Investigator — Paediatric Endocrinology, UKBB
Locations (2):
- Department of Paediatric Endocrinology, Diabetology and Gynaecology, Hôpital Necker-Enfants Malades, Assistance Publique-Hôpitaux de Paris, Paris, France
- Paediatric Endocrinology and Diabetology, University Children's Hospital Basel (UKBB), Basel, Canton of Basel-City, Switzerland